CLINICAL TRIAL: NCT05343650
Title: NOVAPAK Nasal Packing: Safety Study in Shellfish Allergic Patients
Brief Title: NOVAPAK Nasal Packing in Shellfish Allergic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ReDA 12329
Record Dates: First submitted 2022-04-05; First posted 2022-04-25 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Shellfish Hypersensitivity; Epistaxis
Keywords: nasal bleedings; Post-surgical healing; chitosan-based films
MeSH Terms: conditions — Shellfish Hypersensitivity; Epistaxis

STUDY DESIGN:
Intervention Model Description: prospective interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): Stage 1 After shellfish allergy is confirmed through the skin prick test and IgE analysis, Novapak packing will be applied to the patient's skin for 30 minutes on the anterior aspect of the patients' non-dominant arm. In case of pre-existing wounds, it will be applied to the other forearm. Participants will then be monitored for 1 hour, and any- reaction will be documented. In case of any symptoms of an allergic reaction, their study participation will be terminated.
  Stage 2 If no allergic symptoms are observed in stage 1, the patient's nose will be anesthetized with topical lidocaine. A piece of Novapak material will be applied to the participant's nasal cavity at the level of the inferior turbinate for 15 minutes. After removal, the participant will be monitored in the clinic for an hour. Any allergic reaction will be documented, including increased nasal congestion, rhinorrhea, or pruritis.
  Interventions: Device: NOVAPAK nasal packing applied to forearm; Device: NOVAPAK nasal packing applied to nasal cavity

INTERVENTIONS:
Device: NOVAPAK nasal packing applied to forearm — Novapak packing will be applied to the patient's skin for 30 minutes on the anterior aspect of the patients' non-dominant arm. In case of pre-existing wounds, it will be applied to the other forearm.
Device: NOVAPAK nasal packing applied to nasal cavity — A piece of Novapak material will be applied to the participant's nasal cavity at the level of the inferior turbinate for 15 minutes

SUMMARY:
NOVAPAK is a sponge-like material made from materials found in shellfish. It is commonly used after nasal surgery or in nasal bleeding, as it promotes healing, decreases bleeding, and has antibacterial properties. Although NOVOPAK does not contain proteins or compounds known to be responsible for allergic reactions in people with a known allergy to shellfish, out of an abundance of caution, the manufacturer (Medtronic) has recommended avoidance in those with known shellfish allergy. There have been no reported allergic reactions in patients with shellfish allergy who were given chitosan bandages in emergencies (e.g. military applications). The study aims to investigate the safety of its use in patients with known shellfish allergy to improve healthcare quality and patient care support.

DETAILED DESCRIPTION:
This is a prospective interventional study to assess whether the tested product triggers an allergic reaction in patients with known-shellfish allergies.

The primary objective is to assess the safety of Novapak, a chitosan-containing nasal packing material, in patients with known shellfish allergy.

The study will be conducted in two phases. First, participants will undergo an allergy test - Skin prick test (SPT) to crab, lobster, shrimp, oyster, clam, scallop, squid, and octopus -, and antibody levels analysis. Second, in a controlled setting (i.e., in a hospital clinic that includes a resuscitation cart and doctors monitoring - allergist and otolaryngologist), Novapak packing will be applied to the patient's skin for 30 minutes (on the anterior aspect of the patients' non-dominant arm). Then, provided that no allergic symptoms are observed in stage 1, the patient's nose will be anesthetized with topical lidocaine, and a piece of Novapak material will be applied to the participant's nasal cavity at the level of the inferior turbinate for 15 minutes. After removal, the participant will be monitored in the clinic for an hour. Any allergic reaction will be documented, including increased nasal congestion, rhinorrhea, or pruritis.

Since Novapak contains purified chitosan, the investigators hypothesizes that no allergic reactions will be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60
* Positive history of shellfish allergy
* Confirmation of allergy via previous reaction during oral challenge or convincing clinical history and testing.

Exclusion Criteria:

* Severe lung diseases: severe asthma, obstructive lung disease
* Severe cardiovascular disease: history of congestive heart failure, myocardial infarction, valvulopathy, or unstable tachy-or-bradyarrhythmia.
* Severe cerebrovascular disease: history of stroke or severe carotid stenosis.
* Presence of beta-blocker mediations.
* Patients unable to discontinue antihistamine medications or prednisone.
* Patients with severe or refractory anaphylaxis during prior oral challenge to shellfish, or those with documented systemic mastocytosis.
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-12-24 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
First stage - Skin test | Until one hour after the test.
  The occurrence of an Allergic reaction to Novapak packing in the anterior aspect of the patients' non-dominant arm will be tested.
Second stage - Novapak in the nasal cavity (1 hour) | Until one hour after the test
  The occurrence of Allergic reaction to Novapak packing on the participant's nasal cavity at the level of the inferior turbinate.
Second stage - Novapak in the nasal cavity (48 hours) | 48 hours after the test.
  The occurrence of Allergic reaction to Novapak packing on the participant's nasal cavity at the level of the inferior turbinate.

SECONDARY OUTCOMES:
Change in Nasal congestion score - (1 hour) | Baseline, 1 hour after the provocation challenge.
  Change on the nasal congestion score 1 hour after the provocation challenge in the nose using NOVAPAK 0 =No congestion
  1. =Mild congestion
  2. =Moderate congestion
  3. =Severe congestion
Change in Nasal congestion score - (48 hours) | Baseline, 48 hours after the provocation challenge.
  Change on the nasal congestion score 48 hours after the provocation challenge in the nose using NOVAPAK 0 =No congestion
  1. =Mild congestion
  2. =Moderate congestion
  3. =Severe congestion

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurita K. Chitin and chitosan: functional biopolymers from marine crustaceans. Mar Biotechnol (NY). 2006 May-Jun;8(3):203-26. doi: 10.1007/s10126-005-0097-5. Epub 2006 Mar 17. PMID 16532368
- [Background] Chou TC, Fu E, Wu CJ, Yeh JH. Chitosan enhances platelet adhesion and aggregation. Biochem Biophys Res Commun. 2003 Mar 14;302(3):480-3. doi: 10.1016/s0006-291x(03)00173-6. PMID 12615058
- [Background] Rao SB, Sharma CP. Use of chitosan as a biomaterial: studies on its safety and hemostatic potential. J Biomed Mater Res. 1997 Jan;34(1):21-8. doi: 10.1002/(sici)1097-4636(199701)34:13.0.co;2-p. PMID 8978649
- [Background] Winebrake JP, Mahrous A, Kacker A, Tabaee A, Levinger JI, Pearlman AN, Stewart MG, Lelli GJ Jr. Postoperative Bioresorbable Chitosan-Based Dressing for Endoscopic Middle Meatal Dacryocystorhinostomy With Balloon Dilation. Ear Nose Throat J. 2021 Jul;100(6):425-429. doi: 10.1177/0145561319866822. Epub 2019 Sep 26. PMID 31558059
- [Background] Zhou JC, Zhang JJ, Zhang W, Ke ZY, Zhang B. Efficacy of chitosan dressing on endoscopic sinus surgery: a systematic review and meta-analysis. Eur Arch Otorhinolaryngol. 2017 Sep;274(9):3269-3274. doi: 10.1007/s00405-017-4584-x. Epub 2017 Apr 29. PMID 28456847
- [Background] Kourelis K, Shikani AH. Effectiveness of chitosan-based packing in 35 patients with recalcitrant epistaxis in the context of coagulopathy. Clin Otolaryngol. 2012 Aug;37(4):309-13. doi: 10.1111/j.1749-4486.2012.02488.x. No abstract available. PMID 22925096
- [Background] Valentine R, Athanasiadis T, Moratti S, Hanton L, Robinson S, Wormald PJ. The efficacy of a novel chitosan gel on hemostasis and wound healing after endoscopic sinus surgery. Am J Rhinol Allergy. 2010 Jan-Feb;24(1):70-5. doi: 10.2500/ajra.2010.24.3422. PMID 20109331
- [Background] HemCon® Bandage PRO - Tricol Biomedical [Internet]. [cited 2021 Dec 28]. Available from: https://tricolbiomedical.com/product/hemcon-bandage-pro/
- [Background] Waibel KH, Haney B, Moore M, Whisman B, Gomez R. Safety of chitosan bandages in shellfish allergic patients. Mil Med. 2011 Oct;176(10):1153-6. doi: 10.7205/milmed-d-11-00150. PMID 22128651
- [Background] Amaral L, Silva D, Couto M, Nunes C, Rocha SM, Coimbra MA, Coimbra A, Moreira A. Safety of chitosan processed wine in shrimp allergic patients. Ann Allergy Asthma Immunol. 2016 May;116(5):462-3. doi: 10.1016/j.anai.2016.02.004. Epub 2016 Mar 19. No abstract available. PMID 27009439
- [Background] Sicherer SH, Munoz-Furlong A, Sampson HA. Prevalence of seafood allergy in the United States determined by a random telephone survey. J Allergy Clin Immunol. 2004 Jul;114(1):159-65. doi: 10.1016/j.jaci.2004.04.018. PMID 15241360
- [Background] Moonesinghe H, Mackenzie H, Venter C, Kilburn S, Turner P, Weir K, Dean T. Prevalence of fish and shellfish allergy: A systematic review. Ann Allergy Asthma Immunol. 2016 Sep;117(3):264-272.e4. doi: 10.1016/j.anai.2016.07.015. PMID 27613460
- [Background] Lopata AL, Jeebhay MF. Airborne seafood allergens as a cause of occupational allergy and asthma. Curr Allergy Asthma Rep. 2013 Jun;13(3):288-97. doi: 10.1007/s11882-013-0347-y. PMID 23575656
- [Background] Gelis S, Rueda M, Pascal M, Fernandez-Caldas E, Fernandez EA, Araujo-Sanchez G, Bartra J, Valero A. Usefulness of the Nasal Allergen Provocation Test in the Diagnosis of Shellfish Allergy. J Investig Allergol Clin Immunol. 2022 Dec 15;32(6):460-470. doi: 10.18176/jiaci.0736. Epub 2022 Sep 7. PMID 34489219